CLINICAL TRIAL: NCT02841306
Title: Ursodeoxycholic Acid (UDCA) as Adjuvant Treatment for Rhegmatogenous Retinal Detachment: a Phase I Pilot Study
Brief Title: Ursodeoxycholic Acid for Rhegmatogenous Retinal Detachment
Acronym: UDCA-RD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Francine Behar-Cohen (Other)
Collaborators: University of Lausanne Hospitals (Other); Emory University (Other)
Responsible Party: Sponsor-Investigator, Francine Behar-Cohen, Professor, University of Lausanne
Organization: University of Lausanne (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00644
Record Dates: First submitted 2016-07-17; First posted 2016-07-22 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Rhegmatogenous Retinal Detachment
MeSH Terms: interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 3-5 hours (Active Comparator): Duration between oral UDCA intake and surgery of 3-5 hours.
  Interventions: Drug: Ursodeoxycholic Acid
- 6-8 hours (Active Comparator): Duration between oral UDCA intake and surgery of 6-8 hours.
  Interventions: Drug: Ursodeoxycholic Acid
- 9-12 hours (Active Comparator): Duration between oral UDCA intake and surgery of 9-12 hours.
  Interventions: Drug: Ursodeoxycholic Acid
- > 12 hours (Active Comparator): Duration between oral UDCA intake and surgery of >12 hours.
  Interventions: Drug: Ursodeoxycholic Acid
- Control (No Intervention): No medication

INTERVENTIONS:
Drug: Ursodeoxycholic Acid
  Arms: 3-5 hours; 6-8 hours; 9-12 hours; > 12 hours

SUMMARY:
26 patients presenting a rhegmatogenous retinal detachment with more than 4 days of duration will be prospectively included.

A single dose of ursodeoxycholic acid will be administered orally before surgery at different time-points in 22 subjects. Standard surgery will be performed and ocular samples will be collected during the procedure. Ursodeoxycholic acid treatment will be continued in treated patients during 3 months after surgery.

Ocular and serum samples from the 4 untreated patients will serve as negative controls for the determination of UDCA levels.

DETAILED DESCRIPTION:
Retinal detachments consist in a separation of the neuroretina from the retinal pigment epithelium. The most common form is rhegmatogenous retinal detachment (RRD), which occurs as a result of a full-thickness retinal break and the presence of vitreoretinal tractions. Photoreceptor cell death occurs rapidly after RRD and is the ultimate cause of vision loss in these patients. Reattachment of the retina by a surgical procedure allows a recovery of vision. However, the degree of visual recovery differs among patients, despite successful reattachment. This is mainly related to the preoperative visual acuity level, the presence of a macular detachment and its duration. Predicting factors of worse visual acuity are the height of retinal detachment in the macula and the presence of edema, separation, cyst and undulation at the level of the outer nuclear layer showed by optical coherence tomography (OCT). Most patients usually consult with a RRD already involving the macular area after 3 days or more, leading to a worse visual prognostic even with successful surgery. The need for adjuvant neuroprotective agents is then critical to improve photoreceptor survival, functional recovery and subsequent quality of life in patients affected by RRD.

Tauroursodeoxycholic acid (TUDCA) is the taurine conjugate of ursodeoxycholic acid (UDCA), a secondary bile acid produced by intestinal bacteria. UDCA was approved by the Food and Drug Administration (FDA) for the treatment of cholestatic liver disease. Both UDCA and TUDCA are potent inhibitors of apoptosis, in part by interfering with the upstream mitochondrial pathway of cell death, inhibiting oxygen-radical production, reducing endoplasmic reticulum (ER) stress, and stabilizing the unfolded protein response (UPR). TUDCA has been proposed as anti-apoptotic agent in several neurodegenerative diseases, including amyotrophic lateral sclerosis, Alzheimer's, Parkinson's, and Huntington's diseases.

In certain degenerative retinal disorders, such as retinitis pigmentosa, TUDCA plays an important role in preventing cell death. In an animal model of RRD, systemic treatment by TUDCA has been shown to protect photoreceptors from cell death.

The aim of this study is to determine whether detectable levels of UDCA reach the vitreous cavity when administered orally at different time points before surgery for RRD, and to analyze its ocular safety.

20 patients presenting a rhegmatogenous retinal detachment with more than 4 days of duration will be prospectively included.

A single dose of ursodeoxycholic acid will be administered orally before surgery at different time-points in 16 subjects. Standard surgery will be performed and ocular samples will be collected during the procedure. Ursodeoxycholic acid treatment will be continued in treated patients during 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a rhegmatogenous retinal detachment with more than 4 days from symptoms onset.

Exclusion Criteria:

* Previous vitrectomy, vitreous bleeding, other associated retinal disease.
* Monophthalmic patients.
* Pregnancy and lactation, peptic ulcer, acute or chronic liver disease, acute infection of the gallbladder and biliary tract, repeated biliary colic, Crohn's disease, ulcerative colitis, or other disease of the small intestine and colon, and hypersensitivity.
* Patients treated by Cholestyramine, Colestipol and Antacids containing aluminum hydroxide or magnesium, Cyclosporine, Ciprofloxacin, Nitrendipine, Dapsone.
* Patients presenting with galactose intolerance, the Lapp lactase deficiency or glucose and galactose malabsorption.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
UDCA levels in samples from the vitreous | 0-8 months
  concentration in ng/ml

SECONDARY OUTCOMES:
UDCA levels in samples from the sub retinal fluid | 0-8 months
  concentration in ng/ml
UDCA levels in samples from the aqueous humor | 0-8 months
  concentration in ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne, Lausanne, Switzerland